CLINICAL TRIAL: NCT04359784
Title: Phase 2 Pilot Study to Evaluate Efficacy and Safety of Anakinra to Prevent CD19-Targeted CAR-T Cell-Related Cytokine Release Syndrome (CRS) and Neurotoxicity in Patients With B Cell Lymphoma
Brief Title: Anakinra for the Prevention of Cytokine Release Syndrome and Neurotoxicity in Patients With B-Cell Non-Hodgkin Lymphoma Receiving CD19-Targeted CAR-T Cell Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Principal Investigator, Jordan Gauthier, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1006866; NCI-2020-01861 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10373 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6; X-Rays; Phantoms, Imaging; Magnetic Resonance Spectroscopy; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (anakinra, lisocabtagene maraleucel) (Experimental): Patients receive anakinra IV (previously SC) over 10-30 minutes daily on days 0-13 and lisocabtagene maraleucel via infusion on day 0. Patients should also undergo at screening an x-ray, PET/CT or CT, BMA and biopsy (as clinically indicated), and lumbar puncture (as clinically indicated), and at follow-up as clinically indicated. Patients also undergo blood sample collection on study.
  Interventions: Biological: Anakinra; Procedure: X-Ray Imaging; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Lumbar Puncture; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Anakinra — Given IV (previously SC)
  Other Names: Kinaret; Kineret; rIL-1ra; rIL1RN; 143090-92-0
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging; Radiographic Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging; PET scan
Procedure: Computed Tomography — Undergo PET/CT or CT
  Other Names: CAT Scan; Computed Axial Tomography; CT scan
Procedure: Bone Marrow Aspiration — Undergo BMA
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; spinal tap
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase II trial studies how well anakinra works in decreasing the occurrence of cytokine release syndrome (CRS) and damage to the nerves (neurotoxicity) in patients with B-cell non-Hodgkin lymphoma who are receiving CD-19 targeted chimeric antigen receptor T-cell (CAR-T) therapy. CAR-T cell therapy may be complicated by two potentially life-threatening side effects: CRS and neurotoxicity. Anakinra is a drug typically used to treat rheumatoid arthritis, but may also help in preventing CAR-T cell-related cytokine release syndrome and neurotoxicity.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive anakinra intravenously (IV) [previously subcutaneously (SC) for some patients] over 10-30 minutes daily on days 0-13 and lisocabtagene maraleucel via infusion on day 0. Patients should also undergo at screening an x-ray, positron emission tomography/computed tomography (PET/CT) or CT, bone marrow aspirate (BMA) and biopsy (if clinically indicated), and lumbar puncture (if clinically indicated), and at follow-up as clinically indicated. Patients also undergo blood sample collection on study.

After completion of lisocabtagene maraleucel infusion, patients are followed up periodically for up to 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* Karnofsky performance status of >= 60%
* Patients with B-cell non-Hodgkin lymphoma (B-NHL) and eligible for treatment with liso-cel. Patients treated with non-conforming (out-of-specification) liso-cell may remain on study.
* Negative serum pregnancy test within 2 weeks of enrollment for women of childbearing potential, defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year
* Fertile male and female subjects must be willing to use an effective contraceptive method before, during, and for at least 4 months after the last dose of anakinra
* Ability to understand and provide informed consent

Exclusion Criteria:

* Subjects requiring ongoing daily corticosteroid therapy at a dose of > 15 mg of prednisone per day (or equivalent). Pulsed corticosteroid use for disease control is acceptable
* Active autoimmune disease requiring immunosuppressive therapy is excluded unless discussed with the principal investigator (PI)
* Known hypersensitivity to Escherichia € coli-derived proteins, anakinra, or to any component of the product
* Major organ dysfunction defined as:

  * Serum creatinine > 2.5 mg/dL
  * Significant hepatic dysfunction (Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 5x upper limit of normal; bilirubin > 3.0 mg/dL) unless due to malignancy or Gilbert's syndrome in the opinion of the PI or designee
  * Subjects with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing. Those with a forced expiratory volume in 1 second (FEV1) of < 50% of predicted or diffusion capacity of the lung for carbon monoxide (DLCO) (corrected) < 40% will be excluded
  * Significant cardiovascular abnormalities as defined by any one of the following: New York Heart Association (NYHA) class III or IV congestive heart failure, clinically significant hypotension, uncontrolled symptomatic coronary artery disease, or a documented ejection fraction of < 35%
* Uncontrolled serious and active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Gauthier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 27 enrolled participants, 25 met inclusion criteria and started treatment.
Groups:
- Prevention (anakinra, lisocabtagene maraleucel): Participants receive anakinra IV (previously SC) over 10-30 minutes daily on days 0-13 and lisocabtagene maraleucel via infusion on day 0. Participants should also undergo at screening an x-ray, PET/CT or CT, BMA and biopsy (as clinically indicated), and lumbar puncture (as clinically indicated), and at follow-up as clinically indicated. Participants also undergo blood sample collection on study.
  Anakinra: Given IV (previously SC)
  X-Ray Imaging: Undergo x-ray
  Positron Emission Tomography: Undergo PET/CT
  Computed Tomography: Undergo PET/CT or CT
  Bone Marrow Aspiration: Undergo BMA
  Bone Marrow Biopsy: Undergo bone marrow biopsy
  Lumbar Puncture: Undergo lumbar puncture
  Biospecimen Collection: Undergo blood sample collection
Period: Overall Study
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Started | 25
Completed | 23
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Two participants who were enrolled but not treated are included in the baseline analysis population description.
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age Known | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Absence of Any Grade Cytokine Release Syndrome (CRS)
Description: Will assess the efficacy of anakinra in preventing the occurrence of any grade CRS using the Bayesian optimal phase 2 design. Assessed based on the ASTCT Consensus Grading for CRS and Neurotoxicity Associated with Immune Effector Cell.
Time Frame: Up to 28 days after lisocabtagene maraleucel (liso-cel) infusion
Population: Not applicable here (no difference between number of participants analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
Participants
  CRS | 16
  No CRS | 9

2. Secondary Outcome: CRS Grade
Description: CRS severity was graded per American Society for Transplantation and Cellular Therapy (ASTCT) consensus criteria (Lee et al, Biol Blood Marrow Transplant, 2019) based on the presence and severity of fever, hypotension, and hypoxia: grade 1, fever ≥38°C without hypotension or hypoxia; grade 2, hypotension not requiring vasopressors and/or hypoxia requiring low-flow oxygen; grade 3, hypotension requiring a single vasopressor or hypoxia requiring high-flow oxygen; grade 4, life-threatening hypotension requiring multiple vasopressors and/or hypoxia requiring positive-pressure ventilation; grade 5, death.
Time Frame: Up to 28 days after liso-cel infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
Participants
  Peak CRS Grade 0 | 9
  Peak CRS Grade 1 | 8
  Peak CRS Grade 2 | 7
  Peak CRS Grade 3 | 1

3. Secondary Outcome: ICANS Grade
Description: ICANS severity was graded per American Society for Transplantation and Cellular Therapy (ASTCT) consensus criteria (Lee et al, Biol Blood Marrow Transplant, 2019): grade 1, immune effector cell-associated encephalopathy (ICE, overall score range 0-10, higher score = better condition) score 7-9, awakens spontaneously; grade 2, ICE score 3-6, awakens to voice; grade 3, ICE score 0-2, awakens only to tactile stimulus, any clinical seizure that resolves rapidly or non-convulsive seizures on EEG that resolve with intervention, focal/local oedema on neuroimaging; grade 4, ICE 0, unarousable and unable to perform ICE, unarousable or requires vigorous or repetitive tactile stimuli to arouse, stupor or coma, life-threatening prolonged seizure (>5 min); or repetitive clinical or electrical seizures without return to baseline in between, deep focal motor weakness such as hemiparesis or paraparesis, diffuse cerebral oedema on neuroimaging, decerebrate or decorticate posturing, or cranial nerve VI
Time Frame: Up to 28 days after liso-cel infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
Participants
  Peak ICANS Grade 0 | 16
  Peak ICANS Grade 1 | 4
  Peak ICANS Grade 2 | 2
  Peak ICANS Grade 3 | 3

4. Secondary Outcome: Rate of Hospitalization After Liso-cel Treatment
Description: Number of patients hospitalized after liso-cel treatment.
Time Frame: Up to 28 days after liso-cel infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
Participants | 18

5. Secondary Outcome: Duration of Hospitalization After Liso-cel Treatment
Description: Duration of hospitalization measured in days following liso-cel administration.
Time Frame: Up to 28 days after liso-cel infusion
Population: The number of days in the hospital (hospitalized only) group only included patients who were hospitalized (n=18)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
days
  Number of days in the hospital (all pts) | 6 [0 to 10]
  Number of days in the hospital (hospitalized only): number analyzed (Participants) | 18
  Number of days in the hospital (hospitalized only) | 8 [5 to 20]

6. Secondary Outcome: Corticosteroid Usage After Liso-cel Treatment
Description: Number of patients who received corticosteroids within 28 days after liso-cel infusion.
Time Frame: Up to 28 days after liso-cel infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
Participants | 10

7. Secondary Outcome: Disease Response to Liso-cel
Description: Best response within approximately 90 days post liso-cel infusion will be assessed based on institutional standard using physical examination, imaging (CT or PET-CT), and if necessary, bone marrow biopsies, in patients with measurable disease prior to treatment.
Time Frame: Approximately 90 days after liso-cel infusion
Population: Six patients were not evaluable for this endpoint due to lack of measurable disease prior to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
Participants
  CR: number analyzed (Participants) | 19
  CR | 8
  PR: number analyzed (Participants) | 19
  PR | 5
  SD: number analyzed (Participants) | 19
  SD | 2
  PD: number analyzed (Participants) | 19
  PD | 4
  Not evaluable | 6

8. Secondary Outcome: Adverse Events (AEs)
Description: Grade 3 or greater AEs, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 28 days after liso-cel infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed from date of infusion to date off study, up to 32 months; serious adverse events and other (not including serious) adverse events were assessed from the date of consent until stabilization or resolution, up to 36 days after infusion of liso-cel.
Arm/Group | Prevention (anakinra, lisocabtagene maraleucel)
All-Cause Mortality (participants affected / at risk) | 10/25
Serious Adverse Events (participants affected / at risk) | 15/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (anakinra, lisocabtagene maraleucel) (N=25)
Cytokine release syndrome (Immune system disorders) | 11
Fever (General disorders) | 4
Atrial fibrillation (Cardiac disorders) | 2
Chills (General disorders) | 1
Confusion (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Other (Nervous system disorders) | 3 — Immune effector cell-associated neurotoxicity syndrome
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (anakinra, lisocabtagene maraleucel) (N=25)
Lymphocyte count increased (Investigations) | 25
Neutrophil count decreased (Investigations) | 22
White blood cell decreased (Investigations) | 20
Fever (General disorders) | 12
Hypotension (Vascular disorders) | 10
Cytokine release syndrome (Immune system disorders) | 6
Other (Nervous system disorders) | 6 — Immune effector cell-associated neurotoxicity syndrome
Platelet count decreased (Investigations) | 6
Confusion (Psychiatric disorders) | 5
Fatigue (General disorders) | 5
Encephalopathy (Nervous system disorders) | 4
Dysphasia (Nervous system disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Headache (Nervous system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Agitation (Psychiatric disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Chills (General disorders) | 1
Delirium (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fibrinogen decreased (Investigations) | 1
Hallucinations (Psychiatric disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT04359784/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04359784/ICF_000.pdf